CLINICAL TRIAL: NCT06324227
Title: Effects of Multimodal Music Intervention on Cognitive Function, Physical Fitness and Psychology of the Community Dwelling Elderly With Mild Cognitive Impairment
Brief Title: Effects of Multimodal Music Intervention on Mild Cognitive Impairment Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 311203003
Record Dates: First submitted 2024-02-19; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment
Keywords: milc cognitive impairment; cognitive function; music intervention; MMM theory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multimodal music therapy group (Experimental): using twice a week, 12 weeks music intervention with singing and physical movement with rhythm
  Interventions: Other: multimodal music therapy
- no intervention group (Experimental): no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: multimodal music therapy — music therapy
  Arms: multimodal music therapy group
Other: no intervention — no intervention
  Arms: no intervention group

SUMMARY:
The goal of this clinical trial is to learn about whether music therapy can ameliorate cognitive function, physical fitness and psychology in mild cognitive impairment and mild dementia population. The main questions it aims to answer are:

1. To build a model of multimodal music therapy.
2. To discuss the effect of twelve-week multimodal music therapy in ameliorating community-based elders with MCI and mild dementia. Main outcome variables: cognitive function (Montreal Cognitive Assessment Scale, trail making test, Saint Louis University Mental Status Examination). Secondary outcome variables: physical fitness (muscle strength, muscular endurance, flexibility, balance ability), depression.

DETAILED DESCRIPTION:
The prevalence of the elderly with mild cognitive impairment accounts for one-fifth of the elderly population in Taiwan, and there is no medication that can effectively treat the disease. According to the literature review, there are many factors that cognitive impairment would influence. Many chronic diseases can induce cognitive decline, and depression is also related to cognitive function, including memory loss and cognitive decline. Mild cognitive impairment or dementia are also related to disability. Therefore, we choose the music, mood and movement(MMM) theory to connect psychology, cognitive function and physical fitness. The purpose of the research is to establish a model of the multimodal music therapy model and explore the effect of the multimodal music therapy on improving the mild cognitive impairment and mild dementia in the community. The senior with mild cognitive impairment and mild dementia are divided into an experimental group and a control group through randomization consisted of total 49 people based on different day care centers or community-based dementia care centers. It will take 12 weeks for the intervention. The experimental group received multimodal music intervention twice a week, each time with a duration of 70 minutes. The design method partly refers to the methods designed by Shimizu, including three musical instruments for the music therapy and physical activity, and the control group does not have any intervention. The experimental group and the control group have two weeks of pre-test and post-test, and the information sheet of demography, Montreal Cognitive Assessment, Saint Louis University Mental Status Exam, Trail Making Test, muscle strength and endurance, flexibility and dynamic balance ability, Geriatric Depression Scale would be collected before and after the 12-week intervention. The research data is analyzed with Statistical Product and Service Solutions(SPSS). We expect cognitive function, physical fitness and psychology can be improved through multimodal music therapy. This study is also the first time using music, mood and movement theory and applied to multimodal music therapy in Taiwan. If the research results are beneficial, this theory would become a beneficial choice for the elderly with cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with mild dementia
* not diagnosed with dementia, but are suspected cases, including chief complaint or clinical dementia rating scale 0.5.
* more than 65 years old

Exclusion Criteria:

* having severe hearing impairment, or can not talk with Chinese or Taiwanese
* having exercise contraindication
* diagnosed with other psychiatric disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-03-26 (Estimated); Study Completion 2024-05-26 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | about 15 minutes
  The Montreal Cognitive Assessment scale(MoCA) has seven major cognitive functions, including short-term memory, visuospatial, executive function, language ability, attention, abstract reasoning, and orientation. The minimum score is 0 and the highest score is 30. There are total score of 30 points. Considering the literacy, the lower points means the more severe the cognitive function is.
Saint Louis University Mental Status | about 15 minutes
  The Saint Louis University Mental Status(SLUMS) scale includes five major cognitive function: orientation, memory, attention, executive function and language ability. There are 11 questions with a total score of 30 points. The minimum score is 0 and the highest score is 30. There are total score of 30 points. The lower points means the more severe the cognitive function is.
Trail Making Test | about 10 minutes
  The test is designed to examine the attention and can be divided into two parts. There are number 1-25 in circles that appear randomly on the paper. There are Chinese Zodiac and twelve numbers in Trail Making Test-B.

SECONDARY OUTCOMES:
30s chair stand | 30 seconds
  stand up and sit down in 30 seconds to calculate how many times
back scratch test | 15 seconds
  two hands need to reach in your back, one hand on upper and another on lower position
sit and reach test | 15 seconds
  sit on the floor with legs stretched out straight. Then reach forward as far as possible with hands
8-foot up-and-go test | 15 seconds
  calculate the time the participant walk a round trip in a line with 2.44 meters
handgrip | 15 seconds
  participants hold handgrip dynamometer in each hand and squeeze the device as hard as they could to calculate how many kilograms
Geriatric Depression Scale 15 items | 10 minutes
  This 15-question assessment scale is mainly used to detect the tendency of depression in the elderly. Answer "yes" or "no" by reading the questions and comparing their own psychological status. The total score is 0-15. Score 0-4 indicates no tendency to be depressed, 5-10 indicates a tendency to be depressed, and 10-15 indicates a tendency to be severely depressed. The higher the score, the higher the tendency of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Ting Huang, Professor, Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- NationalYangMingU, Taipei, Taiwan